CLINICAL TRIAL: NCT04632641
Title: Suture Closure AFtEr VEIN Access for Cardiac Procedures (SAFE-VEIN) Trial: A Randomized, Prospective Study of the Safety and Efficacy of Venous Closure Device Compared to Conventional Closure Strategies in Post Venous Access Procedures
Brief Title: Suture Closure AFtEr VEIN Access for Cardiac Procedures (SAFE-VEIN) Trial
Acronym: SAFE-VEIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-235
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Heart Block; Pulmonary Embolism and Thrombosis; Mitral Valve Repair; Sinus Node Dysfunction; Bradycardia; Brady-tachy Syndrome
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Heart Block; Pulmonary Embolism; Thrombosis; Sick Sinus Syndrome; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES (Experimental): Perclose ProGlide Suture-Mediated Closure System (SMC) will be used as closure strategy for venous access sites using sheath sizes greater than 13F.
  Interventions: Device: Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES
- Figure 8 Suture - LARGE-BORE PROCEDURES (Active Comparator): Figure 8 suture will be used as a closure technique for venous access sites using sheath sizes greater than 13F.
  Interventions: Other: Figure 8 Suture - LARGE-BORE PROCEDURES

INTERVENTIONS:
Device: Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES — The Perclose ProGlide Suture-Mediated Closure System (SMC) will be used to close the vein access site(s) at the completion of the large-bore procedure in order to achieve hemostasis.
  Arms: Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES
Other: Figure 8 Suture - LARGE-BORE PROCEDURES — A figure 8 suture will be done as a closure strategy in order to achieve hemostasis in large-bore procedures.
  Arms: Figure 8 Suture - LARGE-BORE PROCEDURES

SUMMARY:
Primary objective: To compare the safety and efficacy of closure strategies post venous access procedures.

Hypothesis: We anticipate that the use of a venous closure device will decrease the time to hemostasis (TTH), time to ambulation (TTA) and time to discharge (TTD) compared to conventional methods of closure following venous access procedure.

DETAILED DESCRIPTION:
This study will be a prospective, randomized study of patients who are undergoing one or more of the following procedures at ASLMC (Aurora St. Luke's Medical Center):

Large-Bore Procedures >13 F

1. WATCHMAN® device placement
2. Atrial fibrillation/flutter/SVT (supraventricular tachycardia) ablation using cryoballoon or laser balloon
3. Leadless pacemaker
4. Pulmonary embolism thrombectomy (Inari FlowTriever system)
5. MitraClip transcatheter mitral valve repair

RANDOMIZATION:

Patients will be randomized into one of two venous closure groups after a clean stick has been achieved with no complications:

Large-bore (14F-25F) venous access group (1:1)

* Perclose ProGlide SMC
* Figure 8 suture

ELIGIBILITY:
Inclusion criteria:

Large-bore (>13F) Venous Access Procedures Inclusion Criteria:

All patients 18 years and older who are undergoing any of the following: WATCHMAN® device placement, atrial fibrillation ablation using cryoballoon or laser balloon, leadless pacemaker, Pulmonary embolism thrombectomy (Inari FlowTriever system), MitraClip transcatheter mitral valve repair at Aurora St. Luke's Medical Center from date of IRB (Institutional Review Board) approval through December 2022. All arterial line access should be radial.

Exclusion criteria:

Large-bore (>13F) Venous Access Procedures Exclusion Criteria:

* Patients in whom introducer sheaths >25F were used in the vein during the catheterization procedure.
* Patients with small femoral arteries or veins (< 5 mm in diameter).
* Patients with access sites in vascular grafts.
* Patients with intra-procedural bleeding around access site. Patients who cannot receive radial arterial line access.
* Patients who have complications during the procedure not related to the Perclose ProGlide SMC closure device
* The physician determines that they must use an alternate method as the primary venous closure method other than that which the patient was randomized to
* Active systemic or cutaneous infection, or inflammation in vicinity of the groin
* Pre-existing immunodeficiency disorder or chronic use of high dose systemic steroids
* Known history of bleeding diathesis, coagulopathy, hypercoagulability or platelet count < 100,000 cells/mm3
* Severe co-existing morbidities with life expectancy less than 12 months
* Femoral arteriotomy or femoral venotomy in < 10 days, or with any known vascular complications or residual hematoma, or with use of an intravascular closure device w/in previous 30 days
* Planned femoral venous or arterial access within next 30 days
* Unable to routinely walk at least 20 ft. without assistance
* LMWH (low molecular weight heparin) within 8 hours before or after procedure
* Pregnant and/or lactating women
* Extreme morbid obesity (BMI > 40 kg/m2) or underweight (BMI < 20 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad E Mortada, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Ali M, Masood F, Erickson L, Adefisoye J, Kanani J, Walczak S, Ajam T, Kieu A, Premjee M, Jan MF, Allaqaband SQ, Bajwa T, Khitha J, Zilinski J, Jahangir A, Djelmami-Hani M, Sra J, Niazi I, Mortada ME. Suture closure AFtEr large bore vein access (SAFE-VEIN): A randomized, prospective study of the efficacy and safety of venous closure device. Catheter Cardiovasc Interv. 2024 Oct;104(4):820-828. doi: 10.1002/ccd.31173. Epub 2024 Aug 1. PMID 39087741

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES
Started | 52 | 54
Completed | 47 | 53
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES | Total
Number analyzed (Participants) | 47 | 53 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.5 (10.3) | 69.6 (11.7) | 69.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 27 | 36 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 46 | 53 | 99
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: Kg/m2] | 31.8 (7.1) | 30.3 (6.6) | 31.0 (6.9)
Diabetes Mellitus [Count of Participants; unit: Participants] | 10 | 11 | 21
Hypertension [Count of Participants; unit: Participants] | 27 | 31 | 58
Chronic kidney disease/hemodialysis [Count of Participants; unit: Participants] | 3 | 6 | 9
End stage liver disease [Count of Participants; unit: Participants] | 2 | 0 | 2
Prior stroke or trans ischemic attack [Count of Participants; unit: Participants] | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to Achieve Hemostasis
Description: The elapsed time between "device" removal and first observed and confirmed venous hemostasis
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES
Number analyzed (Participants) | 47 | 53
Minutes | 7 [2 to 10] | 11 [10 to 15]

2. Primary Outcome: Time to Ambulate
Description: The elapsed time between removal of the final Perclose ProGlide SMC device (treatment arm) or removal of the final sheath (control arm), and the ability of subjects to stand and ambulate 20 feet without evidence of venous re-bleeding from the femoral access sites.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES
Number analyzed (Participants) | 46 | 52
Minutes | 322 [246 to 452] | 403 [353 to 633]

3. Secondary Outcome: Time to Discharge (TTD)/Length of Stay (LOS)
Description: The elapsed time between removal of the final sheath, and the ability of subjects to be discharged. Total length of hospital stay.
Time Frame: up to 5 days post procedure
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES
Number analyzed (Participants) | 47 | 53
Minutes | 1257 [1081 to 1544] | 1338 [1171 to 1435]

4. Secondary Outcome: Post Procedure Major Bleeding
Description: Bleeding associated with ≥2 g/dl drop in hemoglobin level requiring transfusion, bleeding that occurs at a critical site, or bleeding contributing to death.
Time Frame: up to 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES
Number analyzed (Participants) | 47 | 53
Participants | 0 | 0

5. Secondary Outcome: Minor Bleeding
Description: Any bleeding that does not meet the criteria for major bleeding
Time Frame: up to 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES
Number analyzed (Participants) | 47 | 53
Participants | 5 | 4

6. Secondary Outcome: Access Site Complications
Description: Access site hematoma, vascular thrombosis, vascular dissection, pseudoaneurysm, or AV (arteriovenous) fistula
Time Frame: up to 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES
Number analyzed (Participants) | 47 | 53
Participants | 0 | 2

7. Secondary Outcome: Mortality
Description: Mortality due to vascular complications
Time Frame: up to 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES
Number analyzed (Participants) | 47 | 53
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Within 30 days of procedure date
Arm/Group | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES | Figure 8 Suture - LARGE-BORE PROCEDURES
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/53
Serious Adverse Events (participants affected / at risk) | 5/47 | 5/53
Other Adverse Events (participants affected / at risk) | 9/47 | 5/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES (N=47) | Figure 8 Suture - LARGE-BORE PROCEDURES (N=53)
GI bleed (Gastrointestinal disorders) | 3 | 0 — Unexpected, unrelated to study
Severe mitral valve regurgitation (Cardiac disorders) | 1 | 0 — Unexpected, unrelated to study
Stroke (Vascular disorders) | 1 | 1 — Unexpected, unrelated to study
Bleeding and Hematoma (Surgical and medical procedures) | 0 | 1 — Expected risk, unrelated to the study
Acute anemia (Blood and lymphatic system disorders) | 0 | 1 — Unexpected, unrelated to study
Oozing (Injury, poisoning and procedural complications) | 0 | 1 — Expected risk, possibly related to the closure method
Bleeding (Injury, poisoning and procedural complications) | 0 | 1 — Expected risk, possibly related to the closure method
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perclose ProGlide Suture-Mediated Closure System (SMC) - LARGE-BORE PROCEDURES (N=47) | Figure 8 Suture - LARGE-BORE PROCEDURES (N=53)
Hematoma (Injury, poisoning and procedural complications) | 0 | 2 — Expected risk, possibly related to study
Bilateral groin bruising/ecchymosis (Injury, poisoning and procedural complications) | 0 | 1 — Expected risk, unlikely related to study
Oozing (Injury, poisoning and procedural complications) | 2 | 0 — Expected risk, possibly related to study
Bleeding (Injury, poisoning and procedural complications) | 2 | 1 — Expected risk, possibly related to study
Hematuria (Renal and urinary disorders) | 2 | 0 — Unexpected risk, unrelated to study
Wrist/forearm pain/swelling and bruising (Injury, poisoning and procedural complications) | 0 | 1 — Unexpected risk, unrelated to study
Atypical chest pain (Cardiac disorders) | 1 | 0 — Unexpected risk, unrelated to study
Chest pain (Infections and infestations) | 1 | 0 — Unexpected risk, unrelated to study
Severe headache and hypertension (General disorders) | 1 | 0 — Unexpected risk, unrelated to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT04632641/Prot_SAP_000.pdf